CLINICAL TRIAL: NCT01461200
Title: A Parallel Group Observational Study of the Effects of Allergic Rhinitis on the Nasal/Sinus Microbiome
Brief Title: Effects of Allergic Rhinitis on the Nasal/Sinus Microbiome
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-712-A
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non allergics
  Interventions: Other: Swab of vestibule and middle meatus of nose
- allergics
  Interventions: Other: Swab of vestibule and middle meatus of nose

INTERVENTIONS:
Other: Swab of vestibule and middle meatus of nose — Swabs of vestibule and middle meatus of nose will be taken prior to and during the grass/tree allergy season

SUMMARY:
The purpose of this study is to find out if the bacteria present in the nose or sinuses of people with seasonal allergies changes during their allergy season. Another purpose of this study is to see if the bacteria present in the nose and sinuses of non-allergic people are the same as allergic people before the allergy season and if it changes during the season. Many bacteria are difficult to grow in the laboratory so the investigators are using analysis of DNA (the genetic material in cells) of the bacteria in the nose and sinus to find them. The investigators will be testing DNA of the bacteria only and not of the human subjects taking part in this study. This research is being done to help us understand how allergy affects bacteria in the nose and sinuses.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 55 years of age.
2. History of tree and/or grass allergic rhinitis for at least 2 years (allergic subjects) or no allergy history at all (normal controls).
3. For allergic subjects, a positive skin test to trees and/or grass antigen within prior 12 months. For non-allergic subjects, negative skin tests to common allergens in the Chicago area.

Exclusion Criteria

1. Respiratory disease other than allergic rhinitis, allergic conjunctivitis and mild asthma.
2. Use of nasal steroids, antihistamines in the last 4 weeks.
3. Upper respiratory infection, sinusitis less than 2 weeks before screening.
4. Structural nasal abnormalities or nasal polyps on examination, nasal ulcer, frequent nose bleeding, recent nasal surgery or nasal trauma (within 90 days).
5. Participation in other investigational therapy in the last 30 days.
6. Any systemic disorder or medication interfering with the study.
7. Undergoing allergen desensitization therapy.
8. Not willing to give informed consent
9. Inability to understand the nature and requirements of the study, or to comply with the study procedures.
10. Any social or medical condition that, in the opinion of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with seasonal allergies and healthy controls from the community.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in bacterial profile of the sinuses | Measured at baseline and 1 to 3 months later.
  DNA isolation to determine the bacterial profiles of samples taken at baseline (out of subjects' allergy season) and 1 to 3 months later during subjects' allergy season.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States